CLINICAL TRIAL: NCT00000312
Title: Alterations in Serotonergic Functions in Cocaine Addicts
Brief Title: Alterations in Serotonergic Functions in Cocaine Addicts - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: NIDA-09468-1; R01-09468-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-12

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — 1-(3-chlorophenyl)piperazine

INTERVENTIONS:
Drug: M-CPP

SUMMARY:
The purpose of this study is to evaluate alterations in the serotonergic system in cocaine addicts and attempt to dissociate changes secondary to cocaine use from those associated with premorbid characteristics.

ELIGIBILITY:
Please contact site for information.

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0

PRIMARY OUTCOMES:
Side effects
Neuroendocrine changes
Psychological changes
Craving

CONTACTS AND LOCATIONS:
Overall Officials: Laure Buydens-Branchey, M.D., Principal Investigator — VA Medical Center
Locations (1):
- VA Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Biological Psychiatry (in press) The. AM. Int. on Addictions (in press)